CLINICAL TRIAL: NCT06642012
Title: Comparing Effectiveness and Cost-effectiveness of Cash Plus Interventions in Preventing Acute Malnutrition in Somalia
Brief Title: Cash Plus Interventions for Prevention of Acute Malnutrition in Children Under 5 and Their Mothers in Somalia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Save the Children (Other); Elrha (Other); Ministry of Health, Somalia (Unknown); UK Foreign, Commonwealth & Development Office (FCDO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00024476; 200011671 (Other Grant/Funding Number: Elrha)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition, Child; Wasting Disease; Stunting; Malnutrition; Malnutrition, Mother
Keywords: Social Behavior Change Communication; Cash Transfer; Humanitarian; Malnutrition; Wasting; Somalia
MeSH Terms: conditions — Child Nutrition Disorders; Wasting Syndrome; Growth Disorders; Malnutrition; Cachexia | interventions — CASP8 and FADD-Like Apoptosis Regulating Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Cash only (Active Comparator): Arm 1 participants received the cash only intervention. Households in this arm received 1 mobile cash transfer per month for 6 months.
  Interventions: Other: Cash only
- Arm 2: Cash + Social Behavior Change Communication (SBCC) (Experimental): Arm 2 participants received the cash + social behavior change communication intervention. Household received 1 mobile cash transfer per month for 6 months but mothers also received an SBCC package that included interpersonal communication (1:1 consultations for mothers), bi-monthly group sessions on key health and nutrition topics, and cooking demonstrations.
  Interventions: Other: Cash + Social Behavior Change Communication
- Arm 3: Cash + top-up cash (Experimental): Arm 3 participants received the cash + top-up cash intervention. Households received 1 mobile cash transfer per month for 6 months, receiving the base cash amount plus an additional cash top-up amount.
  Interventions: Other: Cash + top-up cash

INTERVENTIONS:
Other: Cash only — Households received 1 mobile cash transfer per month for 6 months.
  Arms: Arm 1: Cash only
Other: Cash + Social Behavior Change Communication — Households received 1 mobile cash transfer per month for 6 months but mothers also received an SBCC package that included interpersonal communication (1:1 consultations for mothers), bi-monthly group sessions on key health and nutrition topics, and cooking demonstrations.
  Arms: Arm 2: Cash + Social Behavior Change Communication (SBCC)
Other: Cash + top-up cash — Households received 1 mobile cash transfer per month for 6 months, receiving the base cash amount plus an additional cash top-up amount.
  Arms: Arm 3: Cash + top-up cash

SUMMARY:
This trial studied different combinations of cash assistance to families that live in food insecure areas of Somalia and aimed to understand if this cash assistance provided reduced malnutrition of children and mothers.

DETAILED DESCRIPTION:
This study was a mixed-methods cluster-randomized controlled trial implemented in the Bay and Hiran regions of Somalia to study monthly cash assistance interventions across 3 study arms. The intervention was provided for 6 months and included cash plus social and behavior change communication intervention. The investigators studied which combination of assistance was most effective and cost-effective at reducing and preventing child and maternal malnutrition (wasting, stunting, etc.). Enrolled participants were children under 5 and mothers of children under 5. The investigators collected qualitative, quantitative, and cost data to study the intervention across study arms, household experiences with receiving cash, and household factors related to malnutrition. Quantitative household data and anthropometry was collected at baseline, 3 months, and 6 months. Qualitative data was collected through focus group discussions on health/nutrition topics with mothers and fathers of children under 5 who participated in the study. Cost data was collected in consultation with study and program staff to evaluate the cost-efficiency, cost-effectiveness, and societal costs of the intervention. Investigators also monitored the local markets for food availability and price fluctuations to understand its impact on malnutrition in the communities where the trial was being implemented.

ELIGIBILITY:
Inclusion Criteria for Child Participants:

* Enrolled in Save the Children Cash Plus for Nutrition Program
* Ages 6-59 months at baseline
* Mother is enrolled in the study

Exclusion Criteria for Child Participants:

* Received treatment for wasting at baseline
* Had an episode of severe acute malnutrition in the past 12 months

Inclusion Criteria for Mothers:

* Enrolled in Save the Children Cash Plus for Nutrition Program
* At least 18 years old at baseline
* Have a child that is 6-59 months old at baseline
* Voluntarily willing to participant through signed consent form.

Exclusion Criteria for Mothers:

* Currently receiving treatment for wasting
* Had an episode of severe acute malnutrition in the past 12 months

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3384 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Child Wasting Prevalence | Baseline, 3 months, and 6 months
  Child under 5 wasting prevalence was an aggregate measure of children's nutritional status based on the child's MUAC, weight-for-height z-score (WHZ) measurements, and the present of edema. Using the 2013 WHO guidelines on management of severe acute malnutrition in infants and children, at each study timepoint, children were measured and classified as:
  1. without acute malnutrition (MUAC >= 125 mm and WHZ >= -2 SD and no edema),
  2. with moderate acute malnutrition (115 mm <= MUAC < 124.9 mmm and/or -3<=WHZ<-2 and no edema),
  3. severe acute malnutrition (MUAC < 115 mm and/or WHZ <-3 and/or edema).
  Prevalence was estimated with 95% confidence intervals and changes in prevalence were calculated between baseline, 3 months, and 6 months.
Maternal Wasting Prevalence | Baseline, 3 months, and 6 months
  Aggregate measure of maternal mid-upper arm circumference (MUAC) measured at each time point using standard MUAC tape to the nearest 0.1cm. Mothers were classified as 1) Overweight (MUAC > 300 mm), 2) Normal (300>MUAC>=230mm) or 3) With moderate acute malnutrition (MUAC < 230 mm). Prevalence was estimated with 95% confidence intervals and changes in prevalence were calculated between baseline, 3 months, and 6 months.
Child Mid-Upper Arm Circumference | Baseline, 3 months, and 6 months
  Child mid-upper arm circumference (MUAC) was measured to the nearest 0.1 cm by program staff at each study timepoint using standard MUAC tape.
Child Weight-for-Height | Baseline, 3 months, and 6 months
  Child weight-for-height is an aggregate measure using standard anthropometric measures for weight and height. Child weight was measured to the nearest 0.01 kg using a stand on scale and child height was measured to the nearest 0.1 cm using a wooden length board. Weight-for-height z-scores (WHZ) were calculated using 2006 Word Health Organization child growth standards module in STATA. Weight-for-height compares a child's weight to the weight of a child of the same height and sex from a standard 2006 WHO reference population. This weight-for-height z-score is measured in standard deviations from the median weight for children of the same height and sex. The calculation for Z-score is (X-m)/SD; X is the participant child's weight, m is the median weight for children of the same height and sex in the WHO reference population, and SD is the standard deviation of the weight of the reference population. Z-scores range from -5 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Akseer, PhD, Principal Investigator — Johns Hopkins University; Shelley Walton, MPH, RD, Principal Investigator — Johns Hopkins University; Said Mohamoud, Study Director — Save the Children Somalia; Adam Abdulkadir, Study Director — Save the Children Somalia; Qundeel Khattak, Study Director — Save the Children International
Locations (2):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States
- Save the Children Somalia Office, Mogadishu, Somalia

IPD SHARING:
Plan to Share IPD: No
This data was collected on a vulnerable population linked to a large scale cash assistance program in Somalia. The data may be available upon request with permission from local study investigators.

REFERENCES:
- [Derived] Grounds S, Walton S, Alier KK, Garretson S, Mohamoud SA, Abdiqadir SM, Khattak Q, Nur MA, Mohamoud AM, Ismail MO, Mahat MB, Mohamed AA, Mohamed AA, Tripaldi M, Akseer N. Assessing the correlates of wasting among children under five and their mothers in the Bay and Hiran regions of Somalia. J Glob Health. 2025 Dec 12;15:04308. doi: 10.7189/jogh.15.04308. PMID 41384499
- [Derived] Garretson S, Walton S, Alier KK, Grounds S, Khattak Q, Mohamoud SA, Farah AA, Mohamud FM, Mohamoud AM, Mahdi A, Ismail MO, Mahat MB, Loddo F, Tripaldi M, Akseer N. Analysing concordance between MUAC, MUACZ, and WHZ in diagnosing acute malnutrition among children under five in Somalia. J Glob Health. 2025 Dec 12;15:04258. doi: 10.7189/jogh.15.04258. PMID 41383165